CLINICAL TRIAL: NCT02892942
Title: An Innovative Controlled Ovarian Hyperstimulation (COH) Protocol That Combines Large Oocyte Availability and Physiologic Estrogenic Environment for Good Prognosis In Vitro Fertilization and Embryo Transfer (IVF-ET) Patients
Brief Title: NATural Ovarian Stimulation
Acronym: NATOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: MerckSerono Pharmaceuticals (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150947
Record Dates: First submitted 2016-08-25; First posted 2016-09-08 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Infertility
Keywords: Controlled ovarian hyperstimulation; Estradiol; Embryo implantation; Endometrial receptivity; Fertility preservation
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Background therapy which is the usual COH treatment:
  * Recombinant FSH (Gonal-F®, 225 to 450 IU/d; MerckSerono Pharmaceuticals) from day 2 of their menstrual cycle onward,
  * GnRH antagonist (Cetrotide®, MerckSerono Pharmaceuticals) 0.25 mg/day, S.C., starting on day 6 of Gonal-F®.
  Interventions: Drug: Gonal-F®; Drug: Cetrotide®
- NATOS Group (Experimental): Background therapy which is the usual COH treatment:
  * Recombinant FSH (Gonal-F®, 225 to 450 IU/d; MerckSerono Pharmaceuticals) from day 2 of their menstrual cycle onward,
  * GnRH antagonist (Cetrotide®, MerckSerono Pharmaceuticals) 0.25 mg/day, S.C., starting on day 6 of Gonal-F®.
  GnRH antagonist treatment (Cetrotide®, MerckSerono Pharmaceuticals) will be reinforced and patients will receive 1.5 mg/day (6 ampoules of 0.25 mg), S.C., starting on day 1 (S1) of Gonal-F® treatment until dhCG
  Interventions: Drug: Gonal-F®; Drug: Cetrotide®

INTERVENTIONS:
Drug: Gonal-F® — 225 to 450 IU/d; from day 2 of menstrual cycle onward
Drug: Cetrotide® — 0.25 mg/day, starting on day 6 of Gonal-F®.
Drug: Cetrotide® — 1.5 mg/day (6 ampoules of 0.25 mg), starting on day 1 (S1) of Gonal-F® treatment until dhCG
  Arms: NATOS Group

SUMMARY:
To overcome unsuitable effects of controlled ovarian hyperstimulation (COH )while maintaining large oocyte availability, investigators elaborated an innovative protocol (NATural Ovarian Stimulation) that dissociates E2 production from multiple follicle development.

The purpose of this prospective, randomized trial is to demonstrate that, in a good prognosis IVF-ET population, the physiological E2 environment resulting from NATOS significantly improves IVF-ET outcome when compared to the conventional GnRH antagonist protocol.

DETAILED DESCRIPTION:
Controlled ovarian hyperstimulation (COH) seeks to improve IVF-ET results by increasing per-cycle oocyte and embryo availability. Yet, the coexistence of multiple preovulatory follicles engenders compulsory alterations in the endocrine milieu of the follicular phase. The most evident of them are the extremely high serum estradiol (E2) levels. The 10 to 15-fold increase in E2 levels as a result of COH has been shown to provoke unwanted consequences in both embryo quality and uterine receptivity.

Therefore, investigators elaborated an innovative COH protocol (NATural Ovarian Stimulation) that aimed at dissociating E2 production from multiple follicle development. To obtain this effect, they virtually curtailed endogenous LH production by using GnRH antagonist doses as strong and frequent enough to maintain E2 levels around the physiological range during standard exogenous FSH-only administration. Given that high E2 levels are commonly reached in patients having a normal follicle endowment, NATOS should target this group of good prognosis IVF-ET candidates. Indeed, this new COH approach was first tested in a pilot study that included 15 good prognosis IVF-ET candidates, aged 25-35 years, who volunteered to undergo NATOS. 11 out of 15 patients achieved a pregnancy. These pilot results spurred them to conduct a prospective, randomized trial to demonstrate that, in a good prognosis IVF-ET population, the physiological E2 environment resulting from NATOS significantly improves IVF-ET outcome when compared to the conventional GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* IVF-ET candidates (excluding PGD and oocyte donor);
* Body mass index from 18 to 30 kg/m2;
* Non smokers;
* Regular menstrual cycles (25-35 days);
* Presence of both ovaries;
* Antral follicle count (follicles measuring from 3 to 10 mm in diameter) ranging from 10 to 30 on cycle days 2 to 4;
* Serum AMH levels ranging from 0.5 to 5.0 ng/mL;
* Normal endometrium at ultrasound (US) and/or hysteroscopy;
* Informed consent signed

Exclusion Criteria:

* Iatrogenic ovarian insufficiency (surgery, radiotherapy, chemotherapy);
* Uterine abnormalities as demonstrated by pelvic US and/or hysteroscopy;
* Usual contra-indications for COH (cancer risk, blood coagulation disorders, etc)
* Renal insufficiency

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Live birth obtained after IVF-ET | 1 month post-partum
  Live birth defined as delivery ≥ 22 weeks of amenorrhea

SECONDARY OUTCOMES:
Number of oocytes obtained | At oocyte retrieval (14±8 days after start of treatment)

OTHER OUTCOMES:
Number of embryos obtained | At day 2 of embryo development
Clinical pregnancy | 7 weeks of amenorrhea
  Clinical pregnancy defined as pregnancy with an US-detectable gestational sac at 7 weeks of amenorrhea
Embryo implantation | 7 weeks of amenorrhea
  Embryo implantation defined as the total number of intrauterine gestational sacs divided by the total number of embryos transferred
Miscarriage | Between 7 and 13 weeks of amenorrhea
  Miscarriage defined as a pregnancy loss between 7 and 13 weeks of amenorrhea
"Top" quality embryo | 4 and 5 days after hCG administration
  Embryo data assessed by the number of embryos with adequate morphology
Blastulation | 7 days after hCG administration
  Number of cleaving embryos having reached the blastocyst stage
Adverse events occurring during COH | Within the first 30 days after the start of treatment;
  Presence of ovarian hyperstimulation syndrome (OHSS) +/- severity is measured using OHSS evaluation scale
Gestational age at delivery | 1 month post-partum
Birth weight | 1 month post-partum
Pregnancy complications | 1 month post-partum
  antepartum haemorrhage, placental abruption, hypertensive disorders, and perinatal mortality
Patient's quality of life during COH | At 14 days from start of treatment with cetrotide (plus or minus 8 days)
  Fertiqol modified
Reduced serum E2 levels on dhCG (< 800 pg/mL) | the day of hCG administration
  serum E2 levels will be measured from each blood sample obtained during COH
Serum androgens levels during COH | Within the first 19 days after start of treatment with cetrotide (plus or minus 8 days)
  Serum androgens levels (testosterone, SHBG, androstenedione)

CONTACTS AND LOCATIONS:
Overall Officials: RENATO FANCHIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Antoine Béclère, Clamart, France

IPD SHARING:
Plan to Share IPD: No